CLINICAL TRIAL: NCT02000245
Title: Effects of Sympathy and Touch on Anxiety of Patients Undergoing Fiberoptic Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STAF; 1307-042-504 (Other: Seoul National University Hospital)
Record Dates: First submitted 2013-11-20; First posted 2013-12-04 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Anxiety
Keywords: bronchoscopy; anxiety; touch; sympathy
MeSH Terms: conditions — Anxiety Disorders | interventions — Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- verbal expression for compassion (Active Comparator): verbal expression for compassion
  Interventions: Behavioral: verbal expression for compassion
- verbal expression and touch (Active Comparator): verbal expression and touch
  Interventions: Behavioral: verbal expression for compassion; Behavioral: touch
- control (No Intervention): control

INTERVENTIONS:
Behavioral: verbal expression for compassion — The doctor going to perform bronchoscopy tells a short sentence to a patient. (Hello, I'm Dr.OO. During this test, I will keep an eye on you. Don't worry)
  Arms: verbal expression and touch; verbal expression for compassion
Behavioral: touch — The doctor going to perform bronchoscopy puts a hand on the patient's shoulder
  Arms: verbal expression and touch

SUMMARY:
The purpose of this study is to evaluate the effect of verbal expression of sympathy and touch on anxiety of patients undergoing fiberoptic bronchoscopy

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing diagnostic fiberoptic bronchoscopy
* hospitalized patients

Exclusion Criteria:

* patients who have undergone fiberoptic bronchoscopy
* not hospitalized patients
* cognitive impairment
* refusal to enroll

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
change of visual analogue scale (VAS) for anxiety | baseline (arrival at the test room), and follow-up (at least 10 min after baseline, right before undergoing bronchoscopy

SECONDARY OUTCOMES:
Satisfaction of patients after fiberoptic bronchoscopy | within 6 hours after bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, Principal Investigator — Department of Internal Medicine, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea